CLINICAL TRIAL: NCT01207479
Title: A Multi-Center, Open-Label, Feasibility Study to Assess the Safety and Performance of the VitalaTM Continence Control Device When Worn With SUR FIT Natura® Moldable TechnologyTM Skin Barrier Products Over a 12 Hour Period
Brief Title: Study to Assess the Safety and Performance of The VitalaTM Continence Control Device With Natura Moldable Skin Barriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CC-0196-09-A725
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2013-07

CONDITIONS: Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VitalaTM (Experimental): A 43 day study design has been selected in order to capture meaningful safety and performance data of the Vitala™ device when used with these moldable products.
  Interventions: Device: VitalaTM

INTERVENTIONS:
Device: VitalaTM — A 43 day study design has been selected in order to capture meaningful safety and performance data of the Vitala™ device when used with these moldable products.

SUMMARY:
This is a non-randomized, open-label, multi-center clinical study to be conducted at approximately 5 investigative sites in the US that have expertise in the healthcare management of ostomates. Of the 25 subjects, this study targets a minimum of 15 current moldable users while the remaining users can be non-moldable users if moldable users can not be enrolled.

DETAILED DESCRIPTION:
A Multi-Center, Open-Label, Feasibility Study to Assess the Safety and Performance of the Vitala (TM) Continence Control Device When Worn With SUR FIT Natura® Moldable Technology(TM) Skin Barrier Products Over a 12 Hour Period.

This is a non-randomized, open-label, multi-center clinical study to be conducted at approximately 5 investigative sites in the US that have expertise in the healthcare management of ostomates. Of the 25 subjects, this study targets a minimum of 15 current moldable users while the remaining users can be non-moldable users if moldable users can not be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Is of legal consenting age.
* Is able to read, write, and understand the study, the required procedures, and the study related documentation.
* Has signed the informed consent.
* Has an end colostomy of at least 12 weeks duration with formed or semi-formed effluent.
* Currently uses a SUR-FIT Natura® Moldable skin barrier or is willing to wear SUR-FIT Natura® Moldable Skin Barrier in 45mm or 57mm flange sizes. Enrollment will target as many moldable product users as possible.
* The investigator is relatively sure the subject will be able to wear a SUR-FIT Natura® Moldable Skin Barrier in 45mm or 57mm flange.
* Is willing to remove and replace the skin barrier wafer after three days, or more often if desired.
* Has a stoma that protrudes no more than 2 cm at rest (lying down on back).
* Has demonstrated success in wearing a traditional pouching system. (Investigator judgment)
* Has the ability to do complete self-care.

Exclusion Criteria:

* Has known skin sensitivity to any component of the products being tested.
* Has a skin rating of "L2" or greater according to the SACSTM Rating Scale.
* Is receiving radiation in the area of the pouching system.
* Is receiving chemotherapy other than a stable regimen of maintenance chemotherapy.
* Requires convexity.
* Requires a pouch belt while wearing Vitala™.
* Has participated in a clinical study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety measured by the frequency of adverse events (AEs) relating to the stoma (including GI, and surrounding skin events) and stoma and peristomal vascularity. | 28 Days
  Safety will be assessed by measuring the frequency of adverse events (AEs) relating to the stoma (including GI, and surrounding skin events) and stoma and peristomal vascularity.

SECONDARY OUTCOMES:
Performance (Restoration of Continence) | 28 Days
  Performance will be assessed through the restoration of continence
Performance (Subjective Assessment) | 28 Days
  Performance will be assessed subjectively
Performance (Leakage Rates) | 28 Days
  Performance will be assessed through leakage rates

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, PhD, Study Director — ConvaTec Inc.